CLINICAL TRIAL: NCT02243293
Title: A Randomized, Open-Label, Multicenter Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Co-Administration of ABT-493 and ABT-530 With and Without RBV in Subjects With Chronic Hepatitis C Virus (HCV) Genotypes 2, 3, 4, 5 or 6 Infection (SURVEYOR-II)
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Co-Administration of ABT-493 and ABT-530 With and Without RBV in Subjects With Chronic Hepatitis C Virus (HCV) Genotypes 2, 3, 4, 5 or 6 Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-868; 2014-002927-90 (EudraCT Number)
Record Dates: First submitted 2014-09-04; First posted 2014-09-17 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C; Hepatitis C Virus
Keywords: Hepatitis C Virus (HCV); Hepatitis C; Chronic Hepatitis C; interferon free; Hepatitis C Genotype 2; Hepatitis C Genotype 3; Hepatitis C Genotype 4; Hepatitis C Genotype 5; Hepatitis C Genotype 6
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — glecaprevir; pibrentasvir; Ribavirin; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (22):
- Arm A (Experimental): ABT-493 (300 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD for 12 weeks in HCV genotype 2 (GT2) -infected treatment naïve and treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm B (Experimental): ABT-493 (200 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD for 12 weeks in HCV GT2 -infected treatment naïve and treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm C (Experimental): ABT-493 (200 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD and weight-based ribavirin (RBV) divided twice daily (BID) for 12 weeks in HCV GT2 -infected treatment naïve and treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530; Drug: ribavirin (RBV)
- Arm D (Experimental): ABT-493 (300 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD for 12 weeks in HCV genotype 3 (GT3) -infected treatment naïve and treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm E (Experimental): ABT-493 (200 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD for 12 weeks in HCV GT3 -infected treatment naïve and treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm F (Experimental): ABT-493 (200 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD and weight-based ribavirin (RBV) divided BID for 12 weeks in HCV GT3 -infected treatment naïve and treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530; Drug: ribavirin (RBV)
- Arm G (Experimental): ABT-493 (200 mg) once daily (QD) co-administered with ABT-530 (40 mg) QD for 12 weeks in HCV GT3 -infected treatment naïve and treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm H (Experimental): ABT-493 (200 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD for 8 weeks in HCV GT2 -infected treatment naïve and treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm I (Experimental): ABT-493 (200 mg) once daily (QD) co-administered with ABT-530 (40 mg) QD for 8 weeks in HCV GT2 -infected treatment naïve and treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm J (Experimental): ABT-493 (300 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD for 8 weeks in HCV GT2 -infected treatment naïve and treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm K (Experimental): ABT-493 (200 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD for 8 weeks in HCV GT3 -infected treatment naïve and treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm L (Experimental): ABT-493 (300 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD for 8 weeks in HCV GT3 -infected treatment naïve and for 12 weeks in HCV GT3 -infected treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm M (Experimental): ABT-493 (200 mg) once daily (QD) co-administered with ABT-530 (80 mg) QD for 12 weeks in HCV GT3 -infected treatment naïve participants with compensated cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm N (Experimental): ABT-493 (200 mg) once daily (QD) co-administered with ABT-530 (80 mg) QD and ribavirin (RBV) (800 mg) QD for 12 weeks in HCV GT3 -infected treatment naïve participants with compensated cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530; Drug: ribavirin (RBV)
- Arm O (Experimental): ABT-493 (300 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD for 12 weeks in HCV GT3 -infected treatment naïve participants with compensated cirrhosis and for 16 weeks in HCV GT3 -infected treatment-experienced participants with compensated cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Arm P (Experimental): ABT-493 (300 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD and RBV (800 mg) QD for 12 weeks in HCV GT3-infected treatment naïve and treatment-experienced participants with compensated cirrhosis.
  Interventions: Drug: ABT-493; Drug: ABT-530; Drug: ribavirin (RBV)
- Arm Q1 (Experimental): ABT-493/ ABT-530 (300 mg/ 120mg ) once daily (QD) for 12 weeks in HCV GT3 -infected treatment naïve participants with cirrhosis.
  Interventions: Drug: ABT-493/ABT-530
- Arm Q2 (Experimental): ABT-493/ ABT-530 (300 mg/ 120mg ) once daily (QD) for 12 weeks in HCV GT3 -infected treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493/ABT-530
- Arm R1 (Experimental): ABT-493/ ABT-530 (300 mg/ 120 mg) QD for 16 weeks in HCV GT3 -infected treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493/ABT-530
- Arm R2 (Experimental): ABT-493/ ABT-530 (300 mg/ 120 mg) QD for 16 weeks in HCV GT3 -infected treatment experienced participants with cirrhosis.
  Interventions: Drug: ABT-493/ABT-530
- Arm S1 (Experimental): ABT-493/ ABT-530 (300 mg/ 120 mg) QD for 8 weeks in HCV GT2 infected treatment naïve and treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493/ABT-530
- Arm S2 (Experimental): ABT-493/ ABT-530 (300 mg/ 120 mg) QD for 8 weeks in HCV GT4-6 infected treatment naïve and treatment experienced participants without cirrhosis.
  Interventions: Drug: ABT-493/ABT-530

INTERVENTIONS:
Drug: ABT-493 — Tablet
  Other Names: glecaprevir
  Arms: Arm A; Arm B; Arm C; Arm D; Arm E; Arm F; Arm G; Arm H; Arm I; Arm J; Arm K; Arm L; Arm M; Arm N; Arm O; Arm P
Drug: ABT-530 — Tablet
  Other Names: pibrentasvir
  Arms: Arm A; Arm B; Arm C; Arm D; Arm E; Arm F; Arm G; Arm H; Arm I; Arm J; Arm K; Arm L; Arm M; Arm N; Arm O; Arm P
Drug: ribavirin (RBV) — Tablet
  Arms: Arm C; Arm F; Arm N; Arm P
Drug: ABT-493/ABT-530 — Tablet; ABT-493 co-formulated ABT-530
  Other Names: ABT-493 also known as glecaprevir; ABT-530 also known as pibrentasvir; MAVYRET
  Arms: Arm Q1; Arm Q2; Arm R1; Arm R2; Arm S1; Arm S2

SUMMARY:
The purpose of this phase 2/3, open-label, multipart, multicenter study was to evaluate the efficacy, and safety of co-administration of ABT-493 and ABT-530 with and without ribavirin (RBV) in chronic HCV genotype 2 (GT2-), genotype 3 (GT3-), genotype 4 (GT4), genotype 5 (GT5-), or genotype 6 (GT6-) infected participants with or without cirrhosis.

DETAILED DESCRIPTION:
The study consisted of four independent parts with treatment and post-treatment periods of enrollment. Parts 1 and 2 were the supportive/ exploratory parts (phase 2) of the study and part 3 and 4 were the confirmatory/ registrational parts (phase 3) of the study. In parts 1 and 2 of the study, ABT-493 and ABT-530 were co-administered as separate tablets. However, in parts 3 and 4 of the study, the ABT-493/ABT-530 co-formulated tablets were administered.

ELIGIBILITY:
Inclusion Criteria:

* Screening laboratory result indicating HCV Genotype 2, 3, 4, 5, or 6 infection.
* Chronic HCV infection.
* Participant had to be either HCV treatment-naïve or treatment-experienced.
* Participant had to be documented as non-cirrhotic or as having compensated cirrhosis (GT3 only).

Exclusion Criteria:

* History of severe, life-threatening or other significant sensitivity to any drug.
* Female who was pregnant, planning to become pregnant during the study, or breastfeeding; or male whose partner was pregnant or planning to become pregnant during the study.
* Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol in the opinion of the investigator.
* Positive test result at Screening for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab).
* HCV genotype performed during screening indicating co-infection with more than one HCV genotype.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 694 (Actual)
Dates: Start 2014-09-19; Primary Completion 2016-10-25 (Actual); Study Completion 2017-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

REFERENCES:
- [Background] Kwo PY, Poordad F, Asatryan A, Wang S, Wyles DL, Hassanein T, Felizarta F, Sulkowski MS, Gane E, Maliakkal B, Overcash JS, Gordon SC, Muir AJ, Aguilar H, Agarwal K, Dore GJ, Lin CW, Liu R, Lovell SS, Ng TI, Kort J, Mensa FJ. Glecaprevir and pibrentasvir yield high response rates in patients with HCV genotype 1-6 without cirrhosis. J Hepatol. 2017 Aug;67(2):263-271. doi: 10.1016/j.jhep.2017.03.039. Epub 2017 Apr 13. PMID 28412293
- [Derived] Brown A, Welzel TM, Conway B, Negro F, Brau N, Grebely J, Puoti M, Aghemo A, Kleine H, Pugatch D, Mensa FJ, Chen YJ, Lei Y, Lawitz E, Asselah T. Adherence to pan-genotypic glecaprevir/pibrentasvir and efficacy in HCV-infected patients: A pooled analysis of clinical trials. Liver Int. 2020 Apr;40(4):778-786. doi: 10.1111/liv.14266. Epub 2019 Oct 18. PMID 31568620
- [Derived] Back D, Belperio P, Bondin M, Negro F, Talal AH, Park C, Zhang Z, Pinsky B, Crown E, Mensa FJ, Marra F. Efficacy and safety of glecaprevir/pibrentasvir in patients with chronic HCV infection and psychiatric disorders: An integrated analysis. J Viral Hepat. 2019 Aug;26(8):951-960. doi: 10.1111/jvh.13110. Epub 2019 May 20. PMID 30977945
- [Derived] Gane E, Poordad F, Zadeikis N, Valdes J, Lin CW, Liu W, Asatryan A, Wang S, Stedman C, Greenbloom S, Nguyen T, Elkhashab M, Worns MA, Tran A, Mulkay JP, Setze C, Yu Y, Pilot-Matias T, Porcalla A, Mensa FJ. Safety and Pharmacokinetics of Glecaprevir/Pibrentasvir in Adults With Chronic Genotype 1-6 Hepatitis C Virus Infections and Compensated Liver Disease. Clin Infect Dis. 2019 Oct 30;69(10):1657-1664. doi: 10.1093/cid/ciz022. PMID 30923816
- [Derived] Flamm S, Reddy KR, Zadeikis N, Hassanein T, Bacon BR, Maieron A, Zeuzem S, Bourliere M, Calleja JL, Kosloski MP, Oberoi RK, Lin CW, Yu Y, Lovell S, Semizarov D, Mensa FJ. Efficacy and Pharmacokinetics of Glecaprevir and Pibrentasvir With Concurrent Use of Acid-Reducing Agents in Patients With Chronic HCV Infection. Clin Gastroenterol Hepatol. 2019 Feb;17(3):527-535.e6. doi: 10.1016/j.cgh.2018.07.003. Epub 2018 Sep 10. PMID 30012435
- [Derived] Asselah T, Kowdley KV, Zadeikis N, Wang S, Hassanein T, Horsmans Y, Colombo M, Calinas F, Aguilar H, de Ledinghen V, Mantry PS, Hezode C, Marinho RT, Agarwal K, Nevens F, Elkhashab M, Kort J, Liu R, Ng TI, Krishnan P, Lin CW, Mensa FJ. Efficacy of Glecaprevir/Pibrentasvir for 8 or 12 Weeks in Patients With Hepatitis C Virus Genotype 2, 4, 5, or 6 Infection Without Cirrhosis. Clin Gastroenterol Hepatol. 2018 Mar;16(3):417-426. doi: 10.1016/j.cgh.2017.09.027. Epub 2017 Sep 22. PMID 28951228
- [Derived] Gane E, Poordad F, Wang S, Asatryan A, Kwo PY, Lalezari J, Wyles DL, Hassanein T, Aguilar H, Maliakkal B, Liu R, Lin CW, Ng TI, Kort J, Mensa FJ. High Efficacy of ABT-493 and ABT-530 Treatment in Patients With HCV Genotype 1 or 3 Infection and Compensated Cirrhosis. Gastroenterology. 2016 Oct;151(4):651-659.e1. doi: 10.1053/j.gastro.2016.07.020. Epub 2016 Jul 25. PMID 27456384
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment into arms H, I, K, M and N was not opened by AbbVie.
Pre-assignment Details: Intent-to-treat population: all participants who received at least 1 dose of study drug
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm H | Arm I | Arm J | Arm K | Arm L | Arm M | Arm N | Arm O | Arm P | Arm Q1 | Arm Q2 | Arm R1 | Arm R2 | Arm S1 | Arm S2
Started | 25 | 24 | 25 | 30 | 31 | 31 | 30 | 0 | 0 | 55 | 0 | 53 | 0 | 0 | 28 | 27 | 40 | 22 | 22 | 48 | 145 | 58
Completed | 23 | 23 | 24 | 29 | 30 | 31 | 27 | 0 | 0 | 53 | 0 | 50 | 0 | 0 | 27 | 26 | 37 | 21 | 22 | 47 | 143 | 55
Not Completed | 2 | 1 | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 2 | 3
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 2
Not completed — Enrolled into a Re-treatment Study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but did'nt receive study drug | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received atleast 1 dose of study drug (ITT population)
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm J | Arm L | Arm O | Arm P | Arm Q1 | Arm Q2 | Arm R1 | Arm R2 | Arm S1 | Arm S2 | Total
Number analyzed (Participants) | 25 | 24 | 25 | 30 | 30 | 31 | 30 | 54 | 53 | 28 | 27 | 40 | 22 | 22 | 47 | 145 | 58 | 691
Age, Customized [Number; unit: participants]
  < 65 years | 21 | 21 | 22 | 28 | 29 | 30 | 28 | 44 | 52 | 26 | 24 | 38 | 18 | 19 | 39 | 128 | 49 | 616
  >= 65 years | 4 | 3 | 3 | 2 | 1 | 1 | 2 | 10 | 1 | 2 | 3 | 2 | 4 | 3 | 8 | 17 | 9 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 7 | 11 | 16 | 12 | 15 | 21 | 21 | 13 | 9 | 16 | 8 | 8 | 11 | 84 | 21 | 293
  Male | 16 | 13 | 18 | 19 | 14 | 19 | 15 | 33 | 32 | 15 | 18 | 24 | 14 | 14 | 36 | 61 | 37 | 398
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 4 | 4 | 3 | 5 | 5 | 6 | 2 | 4 | 2 | 9 | 1 | 0 | 4 | 11 | 2 | 65
  Not Hispanic or Latino | 24 | 22 | 21 | 26 | 27 | 26 | 25 | 48 | 51 | 24 | 25 | 31 | 21 | 22 | 43 | 134 | 56 | 626
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: All participants who received at least 1 dose of study drug (ITT population) with evaluable data; participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm J | Arm L | Arm O | Arm P | Arm Q1 | Arm Q2 | Arm R1 | Arm R2 | Arm S1 | Arm S2
Number analyzed (Participants) | 25 | 24 | 25 | 30 | 30 | 31 | 30 | 54 | 53 | 28 | 27 | 40 | 22 | 22 | 47 | 145 | 58
percentage of participants | 96.0 [80.5 to 99.3] | 100.0 [86.2 to 100.0] | 100.0 [86.7 to 100.0] | 93.3 [78.7 to 98.2] | 93.3 [78.7 to 98.2] | 93.5 [79.3 to 98.2] | 83.3 [66.4 to 92.7] | 98.1 [90.2 to 99.7] | 94.3 [84.6 to 98.1] | 96.4 [82.3 to 99.4] | 100.0 [87.5 to 100.0] | 97.5 [87.1 to 99.6] | 90.9 [72.2 to 97.5] | 95.5 [78.2 to 99.2] | 95.7 [85.8 to 98.8] | 97.9 [94.1 to 99.3] | 93.1 [83.6 to 97.3]

2. Primary Outcome: Percentage of Genotype 2 (GT2) Direct-acting Antiviral Agents (DAA)-Naive Participants (in Part 4, Arm S1) With Sustained Virologic Response 12 Weeks Post-treatment (SVR12) as Compared to Historical Control
Description: as for outcome 1
Time Frame: 12 weeks after the last actual dose of study drug
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm S1
Number analyzed (Participants) | 137
percentage of participants | 98.5 [96.5 to 100.0]
Statistical Analysis 1: Comparison: Arm S1; Test type: Non-Inferiority — The non-inferiority of the rate of sustained virologic response at 12 weeks after treatment as compared to historical control (in genotype 2 (GT2) DAA-naive participants in Part 4, arm S) was analyzed; the lower confidence bound of the 2-sided 95% confidence interval (95% CI) for the percentage of participants with sustained virologic response at 12 weeks after treatment must exceed 89% to achieve noninferiority; Percentage of Participants = 98.5, 95% CI 2-sided [96.5 to 100.0] — 95% CI was calculated using the normal approximation to the binomial distribution

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 Weeks Post-treatment (SVR4)
Description: SVR4 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 4 weeks after the last dose of study drug.
Time Frame: 4 weeks after the last actual dose of study drug
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm J | Arm L | Arm O | Arm P | Arm Q1 | Arm Q2 | Arm R1 | Arm R2 | Arm S1 | Arm S2
Number analyzed (Participants) | 25 | 24 | 25 | 30 | 30 | 31 | 30 | 54 | 53 | 28 | 27 | 40 | 22 | 22 | 47 | 145 | 58
percentage of participants | 96.0 [80.5 to 99.3] | 100.0 [86.2 to 100.0] | 100.0 [86.7 to 100.0] | 93.3 [78.7 to 98.2] | 93.3 [78.7 to 98.2] | 93.5 [79.3 to 98.2] | 93.3 [78.7 to 98.2] | 98.1 [90.2 to 99.7] | 96.2 [87.2 to 99.0] | 96.4 [82.3 to 99.4] | 100.0 [87.5 to 100.0] | 97.5 [87.1 to 99.6] | 95.5 [78.2 to 99.2] | 95.5 [78.2 to 99.2] | 95.7 [85.8 to 98.8] | 97.9 [94.1 to 99.3] | 98.3 [90.9 to 99.7]

4. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment; confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during treatment; or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment.
Time Frame: Up to end of treatment (treatment week 8, 12 or 16 depending on arm) or premature discontinuation from treatment
Population: All participants who received at least 1 dose of study drug (ITT population) with evaluable data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm J | Arm L | Arm O | Arm P | Arm Q1 | Arm Q2 | Arm R1 | Arm R2 | Arm S1 | Arm S2
Number analyzed (Participants) | 25 | 24 | 25 | 30 | 30 | 31 | 30 | 54 | 53 | 28 | 27 | 40 | 22 | 22 | 47 | 145 | 58
percentage of participants | 0 [0.0 to 13.3] | 0 [0.0 to 13.8] | 0 [0.0 to 13.3] | 0 [0.0 to 11.4] | 0 [0.0 to 11.4] | 3.2 [0.6 to 16.2] | 3.3 [0.6 to 16.7] | 0 [0.0 to 6.6] | 1.9 [0.3 to 9.9] | 0 [0.0 to 12.1] | 0 [0.0 to 12.5] | 0 [0.0 to 8.8] | 0 [0.0 to 14.9] | 0 [0.0 to 14.9] | 2.1 [0.4 to 11.1] | 0 [0.0 to 2.6] | 0 [0.0 to 6.2]

5. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment, excluding reinfection.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug (ITT population) with evaluable data, completed treatment, and had HCV RNA <LLOQ at the final treatment visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F | Arm G | Arm J | Arm L | Arm O | Arm P | Arm Q1 | Arm Q2 | Arm R1 | Arm R2 | Arm S1 | Arm S2
Number analyzed (Participants) | 24 | 24 | 25 | 29 | 30 | 28 | 28 | 53 | 51 | 28 | 27 | 39 | 22 | 22 | 46 | 144 | 57
percentage of participants | 0.0 [0.0 to 13.8] | 0.0 [0.0 to 13.8] | 0.0 [0.0 to 13.3] | 3.4 [0.6 to 17.2] | 6.7 [1.8 to 21.3] | 0.0 [0.0 to 12.1] | 7.1 [2.0 to 22.6] | 0.0 [0.0 to 6.8] | 2.0 [0.3 to 10.3] | 3.6 [0.6 to 17.7] | 0.0 [0.0 to 12.5] | 0 [0.0 to 9.0] | 9.1 [2.5 to 27.8] | 4.5 [0.8 to 21.8] | 2.2 [0.4 to 11.3] | 1.4 [0.4 to 4.9] | 0 [0.0 to 6.3]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 20 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) or serious adverse event (SAE) with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | ARM A | ARM B | ARM C | ARM D | ARM E | ARM F | ARM G | ARM J | ARM L | ARM O | ARM P | ARM Q1 | ARM Q2 | ARM R1 | ARM R2 | ARM S1 | ARM S2
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/24 | 0/25 | 0/30 | 0/30 | 0/31 | 0/30 | 0/54 | 0/53 | 0/28 | 1/27 | 0/40 | 0/22 | 0/22 | 0/47 | 1/145 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 1/25 | 0/30 | 0/30 | 2/31 | 0/30 | 1/54 | 1/53 | 2/28 | 2/27 | 1/40 | 1/22 | 1/22 | 3/47 | 1/145 | 1/58
Other Adverse Events (participants affected / at risk) | 12/25 | 11/24 | 22/25 | 19/30 | 20/30 | 23/31 | 18/30 | 26/54 | 40/53 | 20/28 | 21/27 | 30/40 | 12/22 | 13/22 | 31/47 | 78/145 | 32/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARM A (N=25) | ARM B (N=24) | ARM C (N=25) | ARM D (N=30) | ARM E (N=30) | ARM F (N=31) | ARM G (N=30) | ARM J (N=54) | ARM L (N=53) | ARM O (N=28) | ARM P (N=27) | ARM Q1 (N=40) | ARM Q2 (N=22) | ARM R1 (N=22) | ARM R2 (N=47) | ARM S1 (N=145) | ARM S2 (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Delusional disorder, unspecified type (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARM A (N=25) | ARM B (N=24) | ARM C (N=25) | ARM D (N=30) | ARM E (N=30) | ARM F (N=31) | ARM G (N=30) | ARM J (N=54) | ARM L (N=53) | ARM O (N=28) | ARM P (N=27) | ARM Q1 (N=40) | ARM Q2 (N=22) | ARM R1 (N=22) | ARM R2 (N=47) | ARM S1 (N=145) | ARM S2 (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3 | 0 | 2 | 2 | 2 | 1 | 2 | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 3 | 3 | 0 | 0 | 1 | 2 | 0 | 1 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 6 | 2 | 1 | 2 | 2 | 4 | 8 | 6 | 1 | 4 | 1 | 2 | 1 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 3 | 4 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 8 | 2 | 6 | 11 | 0 | 5 | 4 | 3 | 7 | 4 | 2 | 2 | 5 | 18 | 5
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 1 | 4 | 2 | 3 | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 2 | 1
Energy increased (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 3 | 10 | 6 | 5 | 12 | 2 | 7 | 15 | 3 | 8 | 5 | 4 | 4 | 16 | 24 | 13
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 3 | 0 | 1 | 2 | 1 | 1 | 3 | 6 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 4 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 5 | 4 | 1 | 1 | 1 | 1 | 4 | 5 | 2 | 3 | 1 | 0 | 2 | 10 | 3
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 7 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 4 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 0 | 2 | 1 | 0 | 2 | 1 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 3 | 1 | 0 | 3 | 4 | 0 | 4 | 0 | 6 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 1 | 1 | 5 | 0 | 0 | 1 | 2 | 4 | 4 | 1 | 0 | 1 | 7 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Headache (Nervous system disorders) | 1 | 3 | 6 | 4 | 3 | 6 | 5 | 6 | 17 | 5 | 9 | 10 | 5 | 4 | 6 | 17 | 11
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 4 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 6 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 4 | 1
Emotional disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 1 | 2 | 3 | 1 | 3 | 5 | 0 | 5 | 1 | 0 | 0 | 3 | 1 | 2
Irritability (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 4 | 0 | 2 | 0 | 0 | 4 | 1 | 0 | 1 | 1 | 2 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 2 | 4 | 0 | 1 | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 3 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 4 | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 4 | 1 | 2 | 1 | 2 | 0 | 1 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 3 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.